CLINICAL TRIAL: NCT04205396
Title: CAREGIVER: An Randomized Clinical Trial (RCT) to Improve the Burden and Distress of Caring for Persons With Decompensated Cirrhosis
Brief Title: CAREGIVER: A Trial to Improve the Burden and Distress of Caring for Persons With Decompensated Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elliot B. Tapper, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00167479
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Caregivers
Keywords: cirrhosis; hepatic encephalopathy; ascites; varices; liver disease; resilience training; expressive writing
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Ascites; Varicose Veins; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Written emotional disclosure (Experimental)
  Interventions: Behavioral: Written emotional disclosure
- Resilience training (Experimental)
  Interventions: Behavioral: Resilience training
- Control arm (Other)
  Interventions: Other: No treatment

INTERVENTIONS:
Behavioral: Written emotional disclosure — Participants will write five stories (days 8, 11, 14, 17 and 20) about an assigned topic relating to their experiences as a caregiver of someone with advanced liver disease. Rules for the exercise will be provided in an instructions page. Additionally, baseline and outcome measures will be completed.
  Arms: Written emotional disclosure
Behavioral: Resilience training — Participants will write three things that went well at the end of their day (before going to sleep), and what was their role in bringing them. These will be done about every three days (days 8, 11, 14, 17 and 20) for 2 weeks at home. Rules for the exercise will be provided in an instructions page. Additionally, baseline and outcome measures will be completed.
  Arms: Resilience training
Other: No treatment — Participants will complete baseline and outcome assessments and no intervention will be conducted.
  Arms: Control arm

SUMMARY:
The goal of this study is to enroll caretakers of patients with decompensated cirrhosis to determine if written emotional disclosure or resilience training interventions reduce distress and burden among primary informal caregivers.

Caretakers that meet eligibility will complete baseline assessments in person, or if necessary, over the phone and be randomized to be in one of three arms of this study. Materials specific to each study arm will be mailed to the caretakers home along with instructions. Overall, the study will take approximately 2 months and a qualitative interview will also be completed around 3-6 months post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* Primary informal caregiver for a patient with a clinical diagnosis of decompensated cirrhosis with either of the following three clinical criteria:

  1. Child-Turcotte Pugh (CTP) Class A/B/C cirrhosis with an all cause hospitalization within the previous 30 days.
  2. CTP Class B or C cirrhosis with one of the following within the prior 6 months from the date of enrollment:

     1. Ascites (requiring paracentesis or diuretics)
     2. Overt Hepatic Encephalopathy (requiring lactulose or rifaximin/flagyl/neomycin)
     3. Spontaneous Bacterial Peritonitis (SBP)
     4. Hepatic Hydrothorax (requiring diuretics or thoracentesis)
     5. Variceal Bleed (with 1 or more recurrences)
  3. Hepatocellular Carcinoma (HCC)

     1. Any Barcelona Clinic Liver Cancer (BCLC) Stage with CTP Class B or C
     2. BCLC Stage C or D with CTP Class A

Exclusion Criteria:

* Non-English speaking
* Unable or unwilling to provide verbal consent
* Severe cognitive impairment
* Caregiver is participating in another interventional study
* Caregiver has used a personal diary within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Change in burden of caregivers measured using the Zarit Burden Interview (ZBI -12) | At baseline and then at 4 week and 8 weeks
  The short form of the ZBI is a validated short 12-item questionnaire measuring perceived burden associated with care giving. Participants rate each item on a 5-point scale ranging from 0 (never) to 4 (nearly always) the range of possible score is 0 (less burden) to 48 (more burden).

SECONDARY OUTCOMES:
Change in Visual Analogue Score (VAS) | At baseline and then at 4 week and 8 weeks
  The VAS is a measure of health related quality of life (HRQOL). It is a scale from 0 to 100 where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Change in Distress Thermometer (DT) | At baseline and then at 4 week and 8 weeks
  This is a single-item self-report measure of distress. The DT is presented as a 10-point scale in a thermometer format and asks to rate how distressed one felt in the previous week from 0 (not distressed) to 10 (extremely distressed).
Change in Caregiver Captivity Index (CCI) | At baseline and then at 4 week and 8 weeks
  A three-item self-report measure of how much (very much, somewhat, just a little, not at all) a caregiver feels like a captive, or being an unwilling or involuntary incumbent of a caregiver role. Scored on a scale of 4-12 with higher scores being worse

OTHER OUTCOMES:
Rate of Healthcare utilization by care recipient | 6 months after randomization
  Number of hospitalizations, number of unscheduled outpatient visits, number of ER visits

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Tapper, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tapper EB, Saleh ZM, Lizza S, Chen X, Nikirk S, Serper M. CAREGIVER Randomized Trial of Two Mindfulness Methods to Improve the Burden and Distress of Caring for Persons with Cirrhosis. Dig Dis Sci. 2023 Sep;68(9):3625-3633. doi: 10.1007/s10620-023-08042-9. Epub 2023 Jul 27. PMID 37498415